CLINICAL TRIAL: NCT00005261
Title: Urinary Kallikrein and Hypertension: A Prospective Study
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1145; R01HL044738 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To determine whether low total urinary kallikrein activity was prospectively associated with new hypertension onset or elevated blood pressures.

DETAILED DESCRIPTION:
BACKGROUND:

Statistical evidence had been found for a dominant major gene segregating in large pedigrees for high urinary kallikrein levels protecting against hypertension which explained 51 percent of the variance of total urinary kallikrein (TUK). In normotensive adult and pediatric pedigree members, low urinary kallikrein activity was associated with a positive family history of hypertension, stroke, and/or coronary disease.

DESIGN NARRATIVE:

The presence of a previously reported dominant major gene inferred from segregation analysis of total urinary kallikrein activity (TUK) in selected pedigrees was verified on already collected frozen urine specimens. Subjects were rescreened to obtain measured nine year follow-up blood pressure data. Individuals were classified by assigned baseline TUK genotype and tested to determine whether low TUK was prospectively associated with new hypertension onset or elevated blood pressures. Because a major gene effect was implicated, available probes for the structural kallikrein gene or other related products regulating kallikrein were tested for genetic linkage to TUK levels. Correlations with over 600 variables measured at baseline in pedigrees and twins were tested to analyze the strong familiality of environment, refine the genetic analyses to better assign genotypes, and detect gene-environment interactions. All baseline variables except kallikrein, aldosterone, and prostaglandin measurements on frozen urine and follow-up blood pressure had already been collected.

TUK may be a marker for a renal, cellular or other physiological abnormality influencing both TUK expression and susceptibility to hypertension. Therefore, the relationship of TUK to urinary aldosterone, prostaglandin E excretion and already measured urinary electrolytes, plasma renin activity, and baseline and reactive blood pressures was determined. Genetic segregation analyses were performed of the urinary variables and other variables closely associated with TUK.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-07; Study Completion 1993-06

REFERENCES:
- [Background] Hunt SC, Wu LL, Slattery ML, Meikle AW, Williams RR. Environmental determinants of urinary kallikrein excretion. Am J Hypertens. 1993 Mar;6(3 Pt 1):226-33. PMID 8466710